CLINICAL TRIAL: NCT00740818
Title: A Pilot Study: Logan Basic Technique and Auxiliary Abdominal Contacts for Reducing Symptomatology of Primary Dysmenorrhea
Brief Title: Logan Basic and Dysmenorrhea
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Patrick Montgomery, DC, Logan College of Chiropractic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SR1120070131
Record Dates: First submitted 2008-08-21; First posted 2008-08-25 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Menstrual Distress (Dysmenorrhea)
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (No Intervention): The patient will lay prone on the adjustment table 5 minutes, the approximate equivalency of a Logan Basic adjustment. Table will be in proper position according to Logan Basic protocol.
  Interventions: Other: No Intervention
- B (Sham Comparator): A thumb contact will be used against the sacrotuberous ligament as opposed to underneath the ligament. Auxiliary contacts will also be sham adjustments; the spine will be contacted but no force applied.
  Interventions: Procedure: Sham Logan Basic Adjustment
- C (Experimental): Logan Basic adjustment, as well as auxiliary and abdominal contacts, based on the Logan Basic protocol.
  Interventions: Procedure: Logan Basic adjustment

INTERVENTIONS:
Other: No Intervention — The patient will lay prone on the adjustment table 5 minutes, the approximate equivalency of a Logan Basic adjustment. Table will be in proper position according to Logan Basic protocol.
  Arms: A
Procedure: Sham Logan Basic Adjustment — A thumb contact will be used against the sacrotuberous ligament as opposed to underneath the ligament. Auxiliary contacts will also be sham adjustments; the spine will be contacted but no force applied.
  Arms: B
Procedure: Logan Basic adjustment — Logan Basic adjustment, as well as auxiliary and abdominal contacts, based on the Logan Basic protocol.
  Arms: C

SUMMARY:
The purpose of this study is to determine the effects of Logan Basic Technique on symptoms of dysmenorrhea.

DETAILED DESCRIPTION:
Dysmenorrhea, also known in the public realm as the dreaded painful period, is a common condition plaguing millions of women. The familiar symptoms of dysmenorrhea include but are not limited to muscle cramping of the lower abdominal muscles, mood swings, breast tenderness, and heavy flow just to name a few. These common complaints can range from a minor annoyance to debilitating. The allopathic model of medicine has offered up several solutions to this problem most women face during their reproductive phase of life. However, even with these options for menstrual discomfort relief, the problem still remains in overwhelming numbers. The rationale of this study is to possibly provide another safer and more effective treatment using protocols of chiropractic medicine.

According to Merck, dysmenorrhea is simplified as pelvic pain during menses. This condition can also be broken down into two forms-primary dysmenorrhea and secondary dysmenorrhea. Primary dysmenorrhea tends to begin in adolescence with the onset of menses. This form is attributed to histological and hormonal changes to the female reproductive system. The symptoms tend to subside with age and pregnancy. Secondary dysmenorrhea is seen to develop in the adult female and is linked to structural anomalies of the pelvic region. Although both of these cause discomfort to several women, the main focus of this study is on treatment of primary dysmenorrhea as treatment of the secondary form involves addressing the underlying structural dysfunction causing the symptoms. This is out of the scope of this study.

Medical treatment of dysmenorrhea involves a few different facets. The first approach is to treat the symptoms of dysmenorrhea with the use of analgesics which is usually the most popular and convenient option. These medications are over-the-counter and are often effective treatment in mild cases. Another option commonly pursued in the medical realm is addressing the hormonal imbalances involved in symptomatology. This is done by prescribing the use of low dose oral contraceptives. This treatment is popular as it provides a convenient preventative measure for pregnancy in addition to symptom relief in some cases. Surgery, an extreme and last resort, involves anywhere from partial to a complete hysterectomy. With partial hysterectomies, there is a higher risk that symptoms will still be present following surgery. However, following a full hysterectomy the patient is subject to the adverse effects of post menopause including but not limited to increased bone loss.

Although effective in the treatment of dysmenorrhea, the medical options can produce adverse effects on the body. Chiropractic treatment offers a mode of care with limited risks and many benefits to the patient. It is the goal of this study to aid in the support of this statement. It has been documented that spinal manipulation using Flexion-Distraction technique combined with Manual Trigger Point therapy has positive results with short-term relief of symptomatology and disability related to chronic pelvic pain syndrome, which is defined as noncyclic pain in the pelvis lasting longer than three months. Although this condition is separate from dysmenorrhea it can provide some insight into symptomatology affecting this region. The Toftness system has also demonstrated significant improvement in subjects suffering from primary dysmenorrhea when compared to those subjects receiving sham adjustments. Gauntt demonstrated the benefits of Logan Basic Technique and Soft Tissue Manipulation in decreasing the symptoms of painful periods. The combination of these treatments establishes "great promise" in intervention of dysmenorrhea. The goal of this new study is to build on Gauntt's work by possibly duplicating these results. This study also aims to explore the efficacy of utilizing auxiliary abdominal contacts in addition to the Logan Basic Protocols.

Logan Basic Methods of adjusting addresses the correction of the base of the spine, the sacrum. By contacting the sacrotuberous ligament on the side of the anteriorly and inferiorly misaligned sacrum, the doctor corrects the said misalignment to help restore proper function to the affected sacroiliac joint. Furthermore, correction of the foundation of the spine, according to Logan Basic Methods, restores optimum function to the entire spine. To increase the efficacy of this procedure, known as the apex contact, one can also utilize auxiliary contacts. Auxiliary contacts are administered during the apex contact. Specifically, auxiliary abdominal contacts address hollow organ spasms. This may be beneficial in addressing the uterine muscle spasms commonly associated with menses.

Logan Basic encompasses a low force adjusting protocol which can be helpful in treatment of all types of patients. This technique is essentially safe for everyone with no known contraindications. However, with any adjusting technique there are adverse reactions to treatment, although usually minor. Patients can experience increased perspiration with their first few adjustments. Following adjustments, the patient can experience pain associated with muscle soreness, which can be treated with the use of cold compresses for twenty minutes on then twenty minutes off for the first 48 hours after treatment. Muscle soreness usually subsides within a day or two and its occurrence decreases with subsequent treatments. Some patients may experience a toxic reaction to treatment that is described as nausea and/or vomiting. This occurs in individuals with increased exposure to drugs and/or a poor diet. However, it is believed that though this reaction has occurred, these patients were in need of this intervention to eliminate toxins from the body.

For this study, a menstrual distress questionnaire will be utilized to objectively analyze subjective complaints of subjects in this study. This method of analyzing symptoms has been used in past studies including Snyder's study on the Toftness system and dysmenorrhea as well as in Gauntt's study on Logan Basic, Soft Tissue Manipulation, and dysmenorrhea. Moos provides an overview of the utilization of this questionnaire. It has been shown to be quite useful in studies with menstrual distress.

Through the exploration of Logan Basic Methods and auxiliary abdominal contacts in the treatment of dysmenorrhea, it is the hope of the investigators to provide some insight into this common condition affecting and disabling women. This investigation aims to build on previous studies showing the efficacy of chiropractic care in the treatment of menstrual distress. Through investigation of primary dysmenorrhea, this study can hopefully assist in opening the scientific community as well as the females of the current society to safer options in treatment of this common condition.

ELIGIBILITY:
Inclusion Criteria:

* Female Logan students, staff, or faculty
* Minimum of 18 years
* No chiropractic adjustments below T12 throughout the duration of the study
* Suffering from primary dysmenorrhea

Exclusion Criteria:

* Pregnancy
* Endometriosis (if known to have)
* Reproductive cancer of any kind
* NSAIDs and/or any other medical or herbal treatments for symptoms of dysmenorrhea. Oral contraception use for this purpose will not be excluded from the study; however, usage will be noted in the final reporting of this study's results.
* Menopause

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-11 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Menstrual Distress Questionnaire | Before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Logan University, College of Chiropractic, Chesterfield, Missouri, United States